CLINICAL TRIAL: NCT03074331
Title: A Phase 3, Open-label Study to Investigate the Efficacy and Safety of Sofosbuvir/Velpatasvir Fixed Dose Combination for 12 Weeks in Subjects With Chronic Hepatitis C Virus (HCV) Infection
Brief Title: Sofosbuvir/Velpatasvir Fixed Dose Combination for 12 Weeks in Adults With Chronic Hepatitis C Virus (HCV) Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-1521
Record Dates: First submitted 2017-02-24; First posted 2017-03-08 (Actual); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SOF/VEL (Experimental): SOF/VEL for 12 weeks
  Interventions: Drug: SOF/VEL

INTERVENTIONS:
Drug: SOF/VEL — 400/100 mg FDC tablet(s) administered orally once daily
  Other Names: Epclusa®; GS-7977/GS-5816

SUMMARY:
The primary objectives of this study are to evaluate the efficacy, safety, and tolerability of treatment with sofosbuvir/velpatasvir (SOF/VEL) fixed-dose combination (FDC) for 12 weeks in adults with chronic hepatitis C virus (HCV) infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent
* HCV RNA detected at screening
* Chronic HCV infection (≥ 6 months) documented by medical history or liver biopsy
* Classification as treatment naïve or treatment experienced. Approximately 20% may be treatment-experienced.
* Cirrhosis determination (approximately 20% may have cirrhosis)
* Females of childbearing potential must have a negative urine pregnancy test at Screening and on Day 1 prior to enrollment.
* Male individuals and female individuals of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception as described in the study protocol
* Lactating females must agree to discontinue nursing before the study drug is administered
* Adults must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments

Key Exclusion Criteria:

* Current or prior history of any of the following:

  * Clinically-significant illness (other than HCV) or any other major medical disorder that may interfere with individual's treatment, assessment or compliance with the protocol
  * Clinical hepatic decompensation (ie, ascites, encephalopathy or variceal hemorrhage)
  * Liver transplantation
  * Hepatocellular carcinoma (HCC) (as determined by appropriate imaging at screening for those with cirrhosis) or current malignancy for which the patient is receiving treatment or which may interfere with individual's treatment, assessment or compliance with the protocol.
* Screening laboratory parameters outside of defined threshold
* Prior exposure to HCV NS5A inhibitor
* Pregnant or nursing female
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Use of any prohibited concomitant medications as described in study protocol
* Known hypersensitivity to VEL, SOF, or formulation excipients

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (16):
- India (16):
  - Seth GS Medical College and KEM hospital, Mumbai, Maharashtra
  - Government Medical College & Super Speciality Hospital, Nagpur, Maharashtra
  - Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, Delhi, New Delhi
  - Global Hospital-Super Speciality & Transpant Centre (A Unite of Centre for Digestive & Kidney Diseases (India) PVT LTD., Mumbai, Parel
  - Post Graduate Institute of Medical Education and Resesarch (PGIMER), Chandigarh, Punjab
  - YRG Care, Chennai, Tamil Nadu
  - VGM Hospital - Institute of Gastroenterology, Coimbatore, Tamil Nadu
  - Gandhi Hospital, Secunderabad, Telangana
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh
  - Department of Hepatology, School of Digestive and Liver Diseases, Kolkata, West Bengal
  - Institute of Digestive and Liver Disease, Guwahati
  - Global Hospitals, Hyderabad
  - Lakeshore Hospital, Kochi
  - Dayanand Medical College & Hospital, Ludhiana
  - Nirmal Hospital, Surat

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in India. The first participant was screened on 23 March 2017. The last study visit occurred on 07 February 2018.
Pre-assignment Details: 170 participants were screened.
Groups:
- SOF/VEL 12 Weeks: Sofosbuvir/velpatasvir (SOL/VEL) (400/100 mg) fixed-dose combination (FDC) tablet orally once daily for 12 weeks
Period: Overall Study
Arm/Group | SOF/VEL 12 Weeks
Started | 130
Completed | 123
Not Completed | 7
Not completed — Enrolled but Not Treated | 1
Not completed — Lost to Follow-up | 5
Not completed — Withdrew Consent | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- SOF/VEL 12 Weeks: SOL/VEL (400/100 mg) FDC tablet orally once daily for 12 weeks
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 128
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 129
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
HCV Genotype [Count of Participants; unit: Participants]
  Genotype 1 | 28
  Genotype 3 | 90
  Genotype 4 | 7
  Genotype 6 | 1
  Indeterminate | 3
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 5.9 (0.96)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 55
  ≥ 800,000 IU/mL | 74

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set included all enrolled participants who took at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 129
percentage of participants | 93.0 [87.2 to 96.8]
Statistical Analysis 1: Comparison: SOF/VEL 12 Weeks; The SVR12 rate was compared to the pre-specified performance goal of 85% by using a two-sided exact one-sample binomial test at the 0.05 significance level; Test type: Superiority; p = 0.009, 2-sided exact 1-sample binomial test

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to Week 12
Population: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 129
percentage of participants | 0

3. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as the following:
  * On Treatment Virologic Failure: HCV RNA persistently ≥ LLOQ through 12 weeks of treatment (nonresponse), or
  * Relapse: HCV RNA ≥ LLOQ at Posttreatment Week 12 having achieved HCV RNA < LLOQ at end of treatment.
Time Frame: Up to Posttreatment Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 129
percentage of participants | 2.3

ADVERSE EVENTS:
Time Frame: Adverse Events: Up to 12 plus 30 days; All-Cause Mortality: Up to Posttreatment Week 12
Description: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Arm/Group | SOF/VEL 12 Weeks
All-Cause Mortality (participants affected / at risk) | 0/129
Serious Adverse Events (participants affected / at risk) | 1/129
Other Adverse Events (participants affected / at risk) | 0/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL 12 Weeks (N=129)
Rectal haemorrhage (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2016-02-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT03074331/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT03074331/SAP_001.pdf